CLINICAL TRIAL: NCT02651428
Title: Phase 3 Prospective, Multicenter, Double-blind, Randomized, Active Control Study to Demonstrate Safety & Effectiveness of Neutrolin in Preventing Catheter-related Bloodstream Infection in Subjects on Hemodialysis for End Stage Renal Disease
Brief Title: Study Assessing Safety & Effectiveness of a Catheter Lock Solution in Dialysis Patients to Prevent Bloodstream Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CorMedix (Industry)
Collaborators: PPD Development, LP (Industry); JMI Laboratories (Industry); Spectra Clinical Research (Other); Davita Clinical Research (Industry); Frenova Renal Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: LOCK-IT-100
Record Dates: First submitted 2016-01-07; First posted 2016-01-11 (Estimated); Results first posted 2021-08-31 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Kidney Failure, Chronic; Catheter-Related Infections
Keywords: Kidney Failure, Chronic; Catheter-Related Infections; Central Venous Catheter
MeSH Terms: conditions — Kidney Failure, Chronic; Catheter-Related Infections | interventions — taurolidine; Citric Acid; Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neutrolin arm (Experimental): Neutrolin: Neutrolin will be added to the central venous catheter after dialysis as a lock solution
  Interventions: Drug: Neutrolin
- Heparin arm (Active Comparator): Heparin: Heparin will be added to the central venous catheter after dialysis as a lock solution
  Interventions: Drug: Heparin

INTERVENTIONS:
Drug: Neutrolin — Neutrolin® will be instilled into central venous HD catheters at the discontinuation of all dialysis sessions and will be withdrawn prior to the initiation of the next dialysis session
  Other Names: 1.35% taurolidine, 3.5% citrate, heparin 1,000 USP Units/mL
  Arms: Neutrolin arm
Drug: Heparin — Heparin will be instilled into central venous HD catheters at the discontinuation of all dialysis sessions and will be withdrawn prior to the initiation of the next dialysis session
  Other Names: Heparin Sodium
  Arms: Heparin arm

SUMMARY:
The purpose of this study is determine safety and effectiveness of Neutrolin, a catheter lock solution, for prevention of central venous catheter associated bloodstream infection in hemodialysis patients.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate the efficacy and safety of Neutrolin® as a catheter lock solution (CLS) on prevention of catheter-related bloodstream infection (CRBSI), and the incidence of treatment-emergent adverse events in subjects receiving hemodialysis (HD) for the treatment of End Stage Renal Disease (ESRD) when compared with heparin 4,000 USP Units/4mL (1,000 USP Units/mL).

This is a randomized, double-blind, active control, parallel-arm, multicenter study. Six hundred and thirty two subjects will be randomized in a 1:1 ratio to receive either Neutrolin® or the active control heparin (Heparin sodium USP 1,000 units/mL, Benzyl alcohol 9.45 mg/mL and Sodium chloride 9.0 mg/mL) as a CLS.

Approximately 632 randomized subjects are planned for this trial. In this study, one-half of the subjects (316 subjects) will receive Neutrolin as a study drug and the other half will receive heparin 4,000 USP Units/4mL (1,000 USP Units/mL) with benzyl alcohol preservative as a comparator. Subjects will be assigned in a 1:1 ratio using permuted blocks without additional stratification for both groups.

The primary objective of this study is to demonstrate the effectiveness of Neutrolin® as a CLS in ESRD subjects undergoing HD treatment using a permanent, cuffed, tunneled silicone or polyurethane HD catheter. The study will evaluate whether Neutrolin® is superior to the active control heparin by documenting the time to CRBSI and consequently delaying the time until the occurrence of CRBSI.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has ESRD and undergoes chronic HD at least two times per week
2. Subject has a HD catheter that has demonstrated the ability to achieve a minimum blood flow of at least 250 mL/min for at least two consecutive dialysis sessions blood flow to enable successful HD
3. The HD catheter is implanted with the tip in a jugular or subclavian vein
4. The subject is not expected to expire within 180 days
5. The subject is likely to require the use of a CVC for at least 90 days
6. The subject (or the legal guardian) understands the nature of the study and provides written informed consent prior to the study enrollment
7. The subject is willing to comply with specified follow-up evaluations and prescribed dialysis therapy and
8. If female and of childbearing potential, the subject must have a negative pregnancy test at the screening visit (i.e., subject is not pregnant); not be lactating; and use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or hormonal contraceptive (oral, implant, ring, patch) for the duration of the study. (NOTE: The subject must have used the chosen method of birth control for at least 1 month/cycle prior to enrollment into the study).

Exclusion Criteria:

1. Subjects who received antibiotics within the last 14 days
2. Visible evidence of compromised skin integrity is present at the catheter exit site or evidence of a catheter exit site infection
3. Subject has received any thrombolytic treatment (i.e., tPA) in their current catheter within 30 days of randomization
4. Fill volume of HD catheter is unknown or cannot be determined
5. Subjects using any type of antimicrobial-coated or heparin-coated catheter
6. Documented chronic bleeding diathesis, active or recurrent bleeding within 1 month prior to randomization
7. Documented history of an atrial thrombus or known hypercoagulable state
8. Subjects with open, non-healing skin ulcers
9. Current requirement for systemic immunosuppression that would increase risk of infection
10. Active malignancy requiring or anticipated to require chemotherapy likely to cause leukopenia and/or immunosuppression
11. Known allergy or absolute contraindication to citrate, taurolidine or heparin or a history of heparin-induced thrombocytopenia
12. Unstable malignancy
13. Cirrhosis with encephalopathy
14. Subject is currently taking another medication with known systemic drug interaction with citrate, taurolidine, or heparin
15. Subject is currently enrolled in another investigational device and/or drug trial or has participated in another investigational device and/or drug trial within 30 days prior to enrollment
16. Subject is anticipated to receive a renal transplant within 90 days (subjects can be on the transplant list, but a subject with a known or anticipated transplant date within the next 90 days should be excluded)
17. Any other medical condition which renders the subject unable to or unlikely to complete the study, or which would interfere with optimal participation in the study or produce significant risk to the subject.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 806 (Actual)
Dates: Start 2015-12; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antony Pfaffle, MD, Study Director — Chief Scientific Officer
Locations (5):
- United States (5):
  - Riverside Nephrology Physicians/Van Buren Dialysis center, Riverside, California
  - North America Research Institute, San Dimas, California
  - North Beach Dialysis Center Inc., Miami Gardens, Florida
  - Lower Manhattan Dialysis Center, New York, New York
  - Diagnostic Clinic of Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Agarwal AK, Crandon J, Hurlburt E, Michaud M, Pfaffle A, Roy-Chaudhury P, Medina C, Conway PT, Hickey EV 3rd. A plain language summary of the LOCK IT-100 study of taurolidine/heparin catheter lock solution and catheter-related bloodstream infection in hemodialysis. Future Microbiol. 2025 Sep;20(13):855-872. doi: 10.1080/17460913.2025.2547498. Epub 2025 Sep 2. PMID 40891537
- [Derived] Agarwal AK, Roy-Chaudhury P, Mounts P, Hurlburt E, Pfaffle A, Poggio EC. Taurolidine/Heparin Lock Solution and Catheter-Related Bloodstream Infection in Hemodialysis: A Randomized, Double-Blind, Active-Control, Phase 3 Study. Clin J Am Soc Nephrol. 2023 Nov 1;18(11):1446-1455. doi: 10.2215/CJN.0000000000000278. Epub 2023 Sep 6. PMID 37678222

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neutrolin Arm | Heparin Arm
Started | 403 | 403
Completed | 359 | 359
Not Completed | 44 | 44

BASELINE CHARACTERISTICS:
Population: All randomized subjects
Groups:
- Total: Total of all reporting groups
Arm/Group | Neutrolin Arm | Heparin Arm | Total
Number analyzed (Participants) | 403 | 403 | 806
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (14.22) | 60.9 (14.39) | 60.9 (14.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 154 | 338
  Male | 219 | 249 | 468
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 5
  Asian | 15 | 18 | 33
  Native Hawaiian or Other Pacific Islander | 10 | 4 | 14
  Black or African American | 126 | 112 | 238
  White | 248 | 262 | 510
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 403 | 403 | 806

OUTCOME MEASURES:

1. Primary Outcome: Presence of a CAC-Adjudicated Catheter-Related Bloodstream Infection (CRBSI) in Subjects Receiving Hemodialysis for the Treatment of End Stage Renal Disease (ESRD): Final Analysis
Description: CRBSI was defined as the same organism grown from at least one positive blood culture from a peripheral site or bloodline sample, or either the arterial or venous catheter hub. The final assessment of CRBSI was determined by a Clinical Adjudication Committee (CAC) who used both clinical documentation and blood culture results in their assessment.
Time Frame: The event time was the number of days from randomization until the occurrence of a CAC-Adjudicated CRBSI or until the subject was censored. The mean participant duration of exposure to study drug was 174 days (range 4-884 days).
Population: Full Analysis Population - all subjects randomized and receiving one or more doses of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Neutrolin Arm | Heparin Arm
Number analyzed (Participants) | 397 | 398
Participants | 9 | 32
Statistical Analysis 1: Comparison: Neutrolin Arm vs Heparin Arm; The null hypothesis was that there was no difference in the survival functions for CRBSI between the two treatments. Based on 80% power to detect a 55% reduction in the risk of CRBSI relative to the control treatment, a 1:1 randomization, a 2-sided log-rank test, one interim analysis using the method of Pocock, and an overall alpha of 0.05, it was determined that 56 CRBSIs would be needed. These are the results of the final analysis; Test type: Superiority; p = 0.0006, Log Rank — The threshold significance level at the interim and final statistical analyses for the primary efficacy endpoint was 0.0294; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.14 to 0.62] — The numerator for the hazard ratio was the estimated hazard for the Neutrolin treatment arm, and the denominator was the estimated hazard for the Heparin treatment arm

2. Secondary Outcome: Participants With a Study Catheter Removal for Any Reason
Description: Analysis of all catheter removals during the study or until the catheter was removed
Time Frame: The event time was the number of days from randomization until catheter removal for any reason or until the subject was censored. The mean participant duration of exposure to study drug was 174 days (range 4-884 days).
Population: Full Analysis Population - all subjects randomized and receiving one or more doses of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Neutrolin Arm | Heparin Arm
Number analyzed (Participants) | 397 | 398
Participants | 236 | 225
Statistical Analysis 1: Comparison: Neutrolin Arm vs Heparin Arm; The null hypothesis was that there was no difference in the time until catheter removal for any reason between the two treatments; Test type: Superiority; p = 0.4161, Log Rank — The threshold for statistical significance was p < 0.05; Hazard Ratio (HR) = 1.08, 95% CI 2-sided [0.90 to 1.29] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Through a participant's study completion. The mean participant duration of exposure to study drug was 174 days (range 4-884 days).
Description: Adverse events were collected for all participants who received study drug, the Full Analysis Population (n=398 Neutrolin, n=399 Heparin). Subjects who did not receive study medication are not included in the adverse event reporting.
Arm/Group | Neutrolin Arm | Heparin Arm
All-Cause Mortality (participants affected / at risk) | 18/398 | 21/399
Serious Adverse Events (participants affected / at risk) | 159/398 | 167/399
Other Adverse Events (participants affected / at risk) | 314/398 | 315/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neutrolin Arm (N=398) | Heparin Arm (N=399)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 2 (2) | 0 (0)
Arteriovenous fistula site infection (Infections and infestations) | 1 (1) | 1 (1)
Arteriovenous graft site infection (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 5 (5) | 7 (7)
Bacterial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2)
Bronchitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 7 (7) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 4 (4) | 0 (0)
Device related infection (Infections and infestations) | 6 (6) | 8 (8)
Device related sepsis (Infections and infestations) | 2 (2) | 4 (4)
Diabetic foot infection (Infections and infestations) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 2 (2)
Endocarditis staphylococcal (Infections and infestations) | 1 (1) | 1 (1)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Gangrene (Infections and infestations) | 3 (3) | 5 (5)
Gastritis viral (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Histoplasmosis (Infections and infestations) | 1 (1) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 1 (1)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 3 (3)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Klebsiella bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Localized infection (Infections and infestations) | 2 (2) | 1 (1)
Necrotizing soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 4 (4) | 4 (4)
Osteomyelitis acute (Infections and infestations) | 0 (0) | 1 (1)
Pancreatic abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 12 (12) | 21 (21)
Pneumonia haemophilus (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0)
Psoas abscess (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 9 (9) | 14 (14)
Septic shock (Infections and infestations) | 5 (5) | 1 (1)
Serratia bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 1 (1) | 4 (4)
Stenotrophomanas infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Viral sepsis (Infections and infestations) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 13 (13)
Angina pectoris (Cardiac disorders) | 5 (5) | 5 (5)
Angina unstable (Cardiac disorders) | 0 (0) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 6 (6)
Atrial tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 5 (5)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure congestive (Cardiac disorders) | 12 (12) | 7 (7)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 1 (1)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 2 (2) | 3 (3)
Coronary artery occlusion (Cardiac disorders) | 2 (2) | 0 (0)
Ischemic cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 3 (3)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 3 (3)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 2 (2)
Pulseless electrical activity (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Failure to thrive (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 14 (14) | 12 (12)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 10 (10) | 8 (8)
Hyperosmolar state (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 6 (6) | 6 (6)
Hypovolemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Lactic acidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 2 (2) | 1 (1)
Angiopathy (Vascular disorders) | 0 (0) | 1 (1)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 2 (2)
Arterial hemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Dry gangrene (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 10 (10)
Hypertensive crisis (Vascular disorders) | 2 (2) | 6 (6)
Hypertensive emergency (Vascular disorders) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 6 (6) | 3 (3)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusive disease (Vascular disorders) | 2 (2) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 1 (1)
Peripheral ischemia (Vascular disorders) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
Steal syndrome (Vascular disorders) | 4 (4) | 1 (1)
Superior vena cava occlusion (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1)
Vasoconstriction (Vascular disorders) | 0 (0) | 1 (1)
Venous stenosis (Vascular disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (9)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colitis ischemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dumping syndrome (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 4 (4) | 6 (6)
Hematemesis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal ischemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal ulcer hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 3 (3) | 0 (0)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (5) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral hemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 4 (4) | 5 (5)
Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 3 (3)
Guillain-Barre syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhage intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Hemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Hyperglycemic seizure (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Hypoxic-ischemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 2 (2) | 2 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 4 (4) | 1 (1)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 2 (2) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anemia postoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Arteriovenous fistula site hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Eschar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrostomy failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incision site hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb surgery (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural hematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Asthenia (General disorders) | 3 (3) | 2 (2)
Chest pain (General disorders) | 1 (1) | 2 (2)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 5 (5) | 2 (2)
Drug withdrawal syndrome (General disorders) | 1 (1) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 5 (5) | 1 (1)
Edema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Hemorrhagic anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Nephrogenic anemia (Blood and lymphatic system disorders) | 3 (3) | 4 (4)
Normocytic anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 3 (3) | 1 (1)
Device malfunction (Product Issues) | 6 (6) | 1 (1)
Thrombosis in device (Product Issues) | 0 (0) | 1 (1)
Biliary diskynesia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 1 (1)
Cholecystitis chronic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hemobilia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Azotemia (Renal and urinary disorders) | 0 (0) | 1 (1)
End stage renal disease (Renal and urinary disorders) | 2 (2) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal hematoma (Renal and urinary disorders) | 1 (1) | 0 (0)
Blood creatinine phosphokinase MB increased (Investigations) | 0 (0) | 1 (1)
Blood culture positive (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction increased (Investigations) | 0 (0) | 1 (1)
Hemoglobin decreased (Investigations) | 1 (1) | 0 (0)
International normalized ration increased (Investigations) | 2 (2) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 2 (2) | 5 (5)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Diabetic foot (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Chronic lymphocytic leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hyperthyroidism secondary (Endocrine disorders) | 0 (0) | 1 (1)
Myxoedema (Endocrine disorders) | 0 (0) | 1 (1)
Blindness cortical (Eye disorders) | 1 (1) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Protein C deficiency (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypogammaglobulinemia (Immune system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Penile swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neutrolin Arm (N=398) | Heparin Arm (N=399)
Bacteremia (Infections and infestations) | 6 (6) | 9 (9)
Bronchitis (Infections and infestations) | 9 (9) | 5 (5)
Cellulitis (Infections and infestations) | 13 (13) | 14 (14)
Device-related infection (Infections and infestations) | 10 (10) | 17 (17)
Nasopharyngitis (Infections and infestations) | 8 (8) | 3 (3)
Osteomyelitis (Infections and infestations) | 8 (8) | 5 (5)
Pneumonia (Infections and infestations) | 18 (18) | 28 (28)
Sepsis (Infections and infestations) | 11 (11) | 21 (21)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 15 (15)
Urinary tract infection (Infections and infestations) | 12 (12) | 15 (15)
Abdominal pain (Gastrointestinal disorders) | 20 (20) | 27 (27)
Constipation (Gastrointestinal disorders) | 18 (18) | 17 (17)
Diarrhea (Gastrointestinal disorders) | 38 (38) | 30 (30)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 6 (6) | 8 (8)
Nausea (Gastrointestinal disorders) | 26 (26) | 43 (43)
Vomiting (Gastrointestinal disorders) | 24 (24) | 31 (31)
Asthenia (General disorders) | 15 (15) | 12 (12)
Catheter site erythema (General disorders) | 7 (7) | 8 (8)
Non-cardiac chest pain (General disorders) | 10 (10) | 4 (4)
Edema peripheral (General disorders) | 9 (9) | 19 (19)
Pain (General disorders) | 7 (7) | 10 (10)
Peripheral swelling (General disorders) | 9 (9) | 9 (9)
Pyrexia (General disorders) | 15 (15) | 24 (24)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 13 (13) | 20 (20)
Fall (Injury, poisoning and procedural complications) | 17 (17) | 17 (17)
Procedural hypotension (Injury, poisoning and procedural complications) | 18 (18) | 18 (18)
Hypertension (Vascular disorders) | 27 (27) | 39 (39)
Hypotension (Vascular disorders) | 35 (35) | 27 (27)
Fluid overload (Metabolism and nutrition disorders) | 26 (26) | 21 (21)
Hyperkalemia (Metabolism and nutrition disorders) | 27 (27) | 26 (26)
Hypoglycemia (Metabolism and nutrition disorders) | 14 (14) | 10 (10)
Device dislocation (Product Issues) | 9 (9) | 5 (5)
Device malfunction (Product Issues) | 68 (68) | 47 (47)
Device occlusion (Product Issues) | 9 (9) | 9 (9)
Thrombosis in device (Product Issues) | 8 (8) | 16 (16)
Cough (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 30 (30)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 (19) | 30 (30)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 10 (10)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 13 (13)
Dizziness (Nervous system disorders) | 22 (22) | 16 (16)
Headache (Nervous system disorders) | 22 (22) | 22 (22)
Syncope (Nervous system disorders) | 10 (10) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 17 (17)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 23 (23) | 36 (36)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 15 (15) | 22 (22)
Acute myocardial infarction (Cardiac disorders) | 6 (6) | 14 (14)
Angina pectoris (Cardiac disorders) | 10 (10) | 8 (8)
Atrial fibrillation (Cardiac disorders) | 7 (7) | 13 (13)
Bradycardia (Cardiac disorders) | 12 (12) | 11 (11)
Cardiac failure congestive (Cardiac disorders) | 16 (16) | 10 (10)
Tachycardia (Cardiac disorders) | 11 (11) | 22 (22)
Skin ulcer (Skin and subcutaneous tissue disorders) | 10 (10) | 4 (4)
Insomnnia (Psychiatric disorders) | 9 (9) | 7 (7)
Mental status changes (Psychiatric disorders) | 9 (9) | 12 (12)
Anemia (Blood and lymphatic system disorders) | 8 (8) | 16 (16)
Nephrogenic anemia (Blood and lymphatic system disorders) | 10 (10) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT02651428/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-29): https://cdn.clinicaltrials.gov/large-docs/28/NCT02651428/SAP_001.pdf